CLINICAL TRIAL: NCT04331132
Title: Tolvaptan add-on Therapy to Overcome Loop Diuretic Resistance in Acute Heart Failure With Renal Dysfunction
Acronym: DR-AHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gia Dinh People Hospital (Other)
Collaborators: Otsuka Pharmaceutical Vietnam (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 92/CN-HĐĐĐ
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-09

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure; worsening renal function; loop diuretic resistance; vasopressin-2 receptor antagonist
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Intervention Model Description: Acute heart failure patients with wet-warm phenotype whose estimated glomerular filtration rates at admission are above 15 and below 60 mL/min/1.73 m2, and cumulative urine output <300 mL in 2 hours after the first dose of intravenous furosemide will be randomly assigned 1:1 to receive a standard care with uptitrating intravenous furosemide alone or a combination therapy with tolvaptan 15mg once daily for 2 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional diuretic group (Placebo Comparator): The conventional furosemide treatment will follow the modified 2019 Position Statement from the ESC Heart Failure Association
  Interventions: Drug: Tolvaptan 15 MG
- Vasopressin-2 antagonist group (Active Comparator): Tolvaptan 15mg once daily for 2 days will be added-on the furosemide strategy based on the modified 2019 Position Statement from the ESC Heart Failure Association
  Interventions: Drug: Tolvaptan 15 MG

INTERVENTIONS:
Drug: Tolvaptan 15 MG — vasopressin-2 receptor antagonist 15mg once daily is added-on to the conventional diuretic strategy
  Other Names: Samsca

SUMMARY:
Renal dysfunction, which comprises 10%-40% of acute heart failure patients (AHF), plays an important role in diuretic resistance mechanism. DR-AHF was designed to demonstrate the effectiveness of early tolvaptan (a vasopressin-2 receptor antagonist) add-on therapy in acute heart failure patients with renal dysfunction and clinical evidence of loop diuretic resistance.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized controlled trial, which will enroll 128 patients hospitalized due to AHF. These patients with wet-warm phenotype whose estimated glomerular filtration rates at admission are above 15 and below 60 mL/min/1.73 m2, and cumulative urine output <300 mL in 2 hours after the first dose of intravenous furosemide will be randomly assigned 1:1 to receive a standard care with uptitrating intravenous furosemide alone or a combination therapy with tolvaptan 15mg once daily for 2 days. The standard furosemide treatment will follow the modified 2019 Position Statement from the ESC Heart Failure Association. The primary endpoint is the cumulative urine output at 48 hour. Key secondary endpoints include the improvement of fractional excretion of sodium at 6 hour, the total dose of furosemide, the changes in the body weights, the net fluid loss, the lessening of diastolic dysfunction parameters on echocardiography, and the incidence of clinically relevant worsening renal function at 48 hour.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital with a primary diagnosis of acute heart failure with wet-warm phenotype
* Cumulative urine volume output < 300ml within 2 hours after the first dose of intravenous furosemide
* eGFR at admission 15-60ml/min/1.73m2

Exclusion Criteria:

* Acute coronary syndrome
* Anuria
* Sepsis
* Consciousness impairment
* Pregnant or breastfeeding women
* Severe valvular heart diseases (severe valvular stenosis or regurgitation)
* Admission sodium level > 140 mEq/L
* Serum total bilirubin > 3 mg/dL
* Serum potassium > 5.5 mmol/L
* Allergy or contraindication for tolvaptan
* Emergency indication for hemodialysis
* Cardiogenic shock or mechanical circulation support

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-26 (Estimated)

PRIMARY OUTCOMES:
Cumulative urine volume output at 48h after randomization | Hour 48
  Urine volume in mL

SECONDARY OUTCOMES:
Cumulative dose of furosemide at 48h after randomization | Hour 48
  Furosemide dose in mg
Symptom of dyspnea by 7-point Likert scale at 24h and 48h after randomization | Hour 24, Hour 48
  3: markedly better, 2: moderately better, 1: minimally better, 0: no change, -1: minimally worse, -2: moderately worse, -3: markedly worse
Changes in body weight at 24h and 48h after randomization | Hour 24, Hour 48
  weight in gram
Incidence of clinically relevant worsening renal function at 24h and 48h after randomization | Hour 24, Hour 48
  An increase in serum creatinine ≥ 0.3 mg/dL within 48 hours accompanying doubling the dose of furosemide according to the diuretic treatment protocol
Changes in serum electrolytes measured at 12h, 24h and 48h after randomization | Hour 12, Hour 24, Hour 48
  Changes in serum sodium (mmol/L), potassium (mmol/L), chloride (mmol/L)
Changes in urine electrolyte excretion at 6h, 24h and 48h | Hour 6, Hour 24, Hour 48
  Increase in sodium (mmol/L), potassium (mmol/L) and chloride (mmol/L) excretion adjusted for urine creatinine (umol/L)
Changes in NT-proBNP at 48h after randomization | Hour 0, Hour 48
  Changes in NT-proBNP (pg/mL)
Changes in mitral e' on echocardiography | Hour 24, Hour 48
  Average of septal e' (cm/s) and lateral e' (cm/s) on tissue doppler imaging in apical 4-chamber view
Changes in E/e' ratio on echocardiography | Hour 24, Hour 48
  The ratio between mitral E (cm/s) and average e' (cm/s)
Changes in left atrial volume on echocardiography | Hour 24, Hour 48
  Average of left atrial volumes (ml) by Simpson's rule in apical 4-chamber and 2-chamber view
Changes in tricuspid regurgitation maximal velocity on echocardiography | Hour 24, Hour 48
  Tricuspid regurgitation maximal velocity (m/s) by continuous wave doppler in apical 4-chamber view
Changes in inferior vena cava maximal diameter on echocardiography | Hour 24, Hour 48
  Inferior vena cava maximal diameter (mm) in subcostal view

CONTACTS AND LOCATIONS:
Overall Officials: Hai H. Nguyen, Ph.D, Study Chair — Cardiology Department
Locations (1):
- Cardiology Department, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Felker GM, Ellison DH, Mullens W, Cox ZL, Testani JM. Diuretic Therapy for Patients With Heart Failure: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Mar 17;75(10):1178-1195. doi: 10.1016/j.jacc.2019.12.059. PMID 32164892
- [Background] Mullens W, Damman K, Harjola VP, Mebazaa A, Brunner-La Rocca HP, Martens P, Testani JM, Tang WHW, Orso F, Rossignol P, Metra M, Filippatos G, Seferovic PM, Ruschitzka F, Coats AJ. The use of diuretics in heart failure with congestion - a position statement from the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2019 Feb;21(2):137-155. doi: 10.1002/ejhf.1369. Epub 2019 Jan 1. PMID 30600580
- [Derived] Minh NG, Hoang HN, Maeda D, Matsue Y. Tolvaptan Add-on Therapy to Overcome Loop Diuretic Resistance in Acute Heart Failure With Renal Dysfunction (DR-AHF): Design and Rationale. Front Cardiovasc Med. 2022 Jan 27;8:783181. doi: 10.3389/fcvm.2021.783181. eCollection 2021. PMID 35155599